CLINICAL TRIAL: NCT02716363
Title: SMart Angioplasty Research Team: A Multi-center, Open Study to Evaluation the Efficacy and Safety of Rotational Atherectomy With Drug Eluting Stent for Calcified LEsion in Korea (SMART-RACE) Trial
Brief Title: Rotational Atherectomy for Calcified lEsion By Smart Angioplasty Research Team (SMART-RACE)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Hyeon-Cheol Gwon, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-06-157
Record Dates: First submitted 2016-03-07; First posted 2016-03-23 (Estimated); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Device : Rotablator (Experimental): We compare in-hospital and long-term efficacy or safety of elective Rotational Atherectomy versus bailout Rotational Atherectomy and low-volume operator versus high-volume operator in patients with severe calcified lesions treated.
  Interventions: Device: Rotational Atherectomy by Rotablator

INTERVENTIONS:
Device: Rotational Atherectomy by Rotablator

SUMMARY:
Current guidelines recommend the use of rotational atherectomy (RA) for preparation of heavily calcified or severely fibrotic lesions that cannot be crossed by a balloon or adequately dilated before planned stenting (bailout situations). RA emerged in the 1990s as one of several tools to treat luminal obstruction via physical removal of plaque. Although initially explored as an alternative to balloon angioplasty, RA has shown favorable acute results in facilitating stent delivery and adequate expansion, particularly those affected by heavy calcification.Drug-eluting stents (DES) have substantially reduced re-stenosis rates in randomized clinical trials evaluating simple de novo coronary artery lesions and have also shown favorable results when implanted in complex lesions and patients, but higher event rates are observed when treating such subsets compared with simple lesions even with newer generation DES. However, there are limited data on evaluating the safety and effectiveness of RA followed by DES implantation for heavily calcified lesions in contemporary practice. Recent randomized controlled trial shows that RA before paclitaxel eluting stent implantation as first generation DES was not superior to paclitaxel eluting stent implantation without prior RA in reducing the primary endpoint of in-stent late luminal loss at 9 months, indicating that RA does not increase the efficacy of DES in patients with moderate to severe calcified lesions. However, there were only 15 (12.5%) crossovers from standard therapy to rotablation because of failure of balloon or stent delivery or suboptimal balloon expansion despite the use of a noncompliant balloon. Accordingly, procedural and fluoroscopy times were longer in the elective RA and procedural complications occurred equally in both elective RA and bailout RA. These findings might cause by a substantial portion of enrolled population have moderate calcified lesions, but not severe calcified lesions. In particular, everolimus-eluting stent (EES) as newer generation DES could act synergistically in heavily calcified lesions as RA could avert stent coating damage and EES could effectively suppress neointimal proliferation. Therefore, we compare in-hospital and long-term efficacy or safety of elective RA versus bailout RA and low-volume operator versus high-volume operator in patients with severe calcified lesions treated with EES.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 19 years of age
* Angiographically proven coronary artery disease
* Patients underwent Rotational Atherectomy
* He/she or his/her legally authorized representative provides written informed consent
* Target lesion(s) must be located in a native coronary artery with visually estimated diameter of ≥ 2.25 mm and ≤ 4.25 mm

Exclusion Criteria:

* Cardiac arrest before the procedure
* Pregnancy or breast feeding
* Thrombotic lesion
* Saphenous vein graft
* Unprotected left main lesion

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2015-11-01; Primary Completion 2020-08-31 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
A composite procedure-related complication | 2 years
  cardiac death, peri-procedural myocardial infarction (CK-MB rise > X10 URL), coronary perforation, cardiopulmonary resuscitation, hemodynamic support (IABP, PCPS), or emergency surgery

SECONDARY OUTCOMES:
Procedure duration | from guiding catheter to final angiography, an average of 1 day
Fluoroscopy time | from guiding catheter to final angiography, an average of 1 day
Target vessel failure | 1,6 and 12months
  Defined as a composite of cardiac death, myocardial infarction , or target vessel revascularization
Final in-stent minimal lumen area by IntraVascular UltraSound | 1,6 and 12months

CONTACTS AND LOCATIONS:
Locations (1):
- Hyoen-Cheol Gwon, MD,PhD, Seoul, South Korea